CLINICAL TRIAL: NCT05856799
Title: Danish Randomized Trial on VDD Leadless Atrial Tracking With MicraTM AV Transcatheter Pacing System vs Transvenous DDD Pacing in Elderly Patients With AV-block
Brief Title: Danish Randomized Trial on Leadless vs Transvenous Pacing
Acronym: DANVERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DANVERS2303101
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-11

CONDITIONS: AV Block
Keywords: Leadless Pacing; Cardiac Pacemaker; Cardiac Arrythmia; Heart Disease
MeSH Terms: conditions — Atrioventricular Block; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Combined parallel and crossover randomized trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Partly patient and accessor blinded and partly open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leadless Pacemaker (Active Comparator): Implantation with a leadless pacemaker
  Interventions: Device: Leadless Micra AV Transcatheter Pacing System
- Transvenous pacemaker (Active Comparator): Implantation with a transvenous pacemaker
  Interventions: Device: Transvenous Azure XT DR dual chamber pacemaker

INTERVENTIONS:
Device: Leadless Micra AV Transcatheter Pacing System — Patients are implanted with a leadless Micra AV TPS
  Arms: Leadless Pacemaker
Device: Transvenous Azure XT DR dual chamber pacemaker — Patients are implanted with a transvenous Azure XT DR pacemaker
  Arms: Transvenous pacemaker

SUMMARY:
The purpose of this study is to evaluate the quality of life, patient acceptance and exercise capacity with leadless compared to transvenous pacing in elderly patients with new-onset high-grade atrioventricular block. Consecutive patients with high-grade atrioventricular black and preserved sinus node function with indication for permanent pacemaker implantation according to the latest european guidelines, are included in a prospective, partly patient and accessor blinded and partly open label, 1:1 randomized combined parallel and cross-over trial to implantation with 1) a Micra AV Transcathter Pacing System or 2) an Azure XT DR dual chamber pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* First time pacemaker implantation on class I or II ESC recommendations for AVB with an expected amount of right ventricular pacing >80% of the time,
* Age 75 years or older
* Intact sinus node function
* Expected survival more than 12 months based on clinical evaluation
* Able to provide informed consent

Exclusion criteria:

* Persistent or previous cardiac implantable electronic device i.e., pacemaker, ICD, or CRT.
* Persistent, or chronic atrial fibrillation
* Reversible AVB
* Transient AVB due to ongoing ischemia
* Heart failure NYHA class III-IV
* Heart failure with branch block and indication for CRT implantation, irrespective of NYHA class
* Indication for primary or secondary prophylactic ICD implantation
* Acute myocardial infarction (AMI) within 3 months
* Severe chronic pulmonary disease with pulmonal hypertension limiting exercise capacity
* Expected survival < 12 months based on clinical evaluation
* Performing high intensity sport
* Participation in another trial with experimental treatment
* Contraindication against device implantation (e.g., concurrent infection)
* Failure to provide informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Life by SF36 | 7 months
  Self-reported health-related quality of life as measured by Short-Form 36 quality of life questionnaire. The scale ranges from 0 to 100. 0 denotes minimal quality of life and 100 denotes maximum quality of life.

SECONDARY OUTCOMES:
Patient Acceptance by FPAS | 7 months
  Self-reported patient acceptance as measured by Florida Patient Acceptance Scale. The scale ranges from 0-100. 0 denotes minimal device acceptance and 100 denotes maximal device acceptance.
Exercise capacity by 6MWT | 7 months
  Exercise capacity as measured by 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Mads B. Kronborg, DMSc, Principal Investigator — Department of Cardiology Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Cardiology Aarhus University Hospital, Aarhus, Region Midt
  - Department of Cardiology Odense University Hospital, Odense, Region Syd

IPD SHARING:
Plan to Share IPD: No
In accordance with Danish and European data protection law